CLINICAL TRIAL: NCT05545657
Title: A Cross-sectional and Longitudinal Study to Investigate the Relationship and Central Mechanism Between Diabetes and Cognitive Impairment Based on Simultaneous EEG-fMRI Approach and Peripheral Neuropathology Biomarkers Assay
Brief Title: Relationship and Central Mechanism Between Diabetes and Cognitive Impairment Based on Simultaneous EEG-fMRI Approach and Peripheral Neuropathology Biomarkers Assay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-MS-03
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes; Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: These patients must have a definite diagnosis of type 2 diabetes mellitus (T2DM) according to the American Diabetes Association (ADA) standards. Some of these patients have symptoms of cognitive impairment, while others have normal cognition.
  Interventions: Behavioral: Cognitive assessments; Other: Simultaneous EEG-fMRI scan; Other: Multimodal magnetic resonance imaging; Other: Peripheral blood neuropathology biomarkers assay
- Healthy Control: These participants have normal glucose tolerance and normal cognition.
  Interventions: Behavioral: Cognitive assessments; Other: Simultaneous EEG-fMRI scan; Other: Multimodal magnetic resonance imaging; Other: Peripheral blood neuropathology biomarkers assay

INTERVENTIONS:
Behavioral: Cognitive assessments — Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Rey Auditory Verbal Learning Test (RAVLT), Boston Naming Test (BNT), Digit Span Test (DST), Trail Making Test (TMT).
Other: Simultaneous EEG-fMRI scan — EEG recordings were conducted with a 64-channel MR-compatible EEG system (Electrical Geodesics Inc., Eugene, OR, USA) and an MR-compatible EEG cap (HydroCel Geodesic Sensor Nets), using ring-type sintered silver chloride electrodes with iron-free copper leads.
Other: Multimodal magnetic resonance imaging — 3D T1-weighted imaging, Resting-state fMRI, Diffusion tensor imaging, Arterial spin labeling.
Other: Peripheral blood neuropathology biomarkers assay — Detecting the peripheral blood neuropathology biomarkers using single molecule array (Simoa) technique, including Aβ40, Aβ42, P-tau 181, P-tau 231, GFAP and NfL.

SUMMARY:
This is a cross-sectional and longitudinal study to investigate the relationship and central mechanism between type 2 diabetes and cognitive impairment based on the simultaneous EEG-fMRI approach and peripheral neuropathology biomarkers assay.

DETAILED DESCRIPTION:
Little is known about the high risks of cognitive impairment and Alzheimer's Disease (AD) in people with type 2 diabetes. The goal of this study is to characterize brain imaging biomarkers of preclinical AD and related cognitive impairment in people with type 2 diabetes using the simultaneous EEG-fMRI approach and peripheral neuropathology biomarkers assay. We will recruit 400 patients with type 2 diabetes in the outpatient and inpatient departments. Each subject will undergo simultaneous EEG-fMRI scan, classical multimodal MRI scan, cognitive assessments and peripheral neuropathology biomarkers assay at the baseline. This study will qualify gray matter volume, cortical thickness, gray matter and white matter microstructure, cerebral blood flow, spectrum changes, as well as resting state and dynamic functional network connectivity from the imaging examination. Study duration was 3 years with a follow-up every 12 months. Cognitive assessments and imaging scan will be conducted in each follow-up visits. At the end of the study, all of the assessments will be performed again for all recruited subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-75 years
* Right handedness
* Possessed over 6-year education
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* Control participants would be excluded if they had a fasting blood glucose level >7.0 mmol/L; glucose level> 7.8 mmol/L after oral glucose tolerance test (OGTT); HbA1c>5.7%
* Control participants would be excluded if they had a Montreal Cognitive Assessment (MoCA, Beijing edition) score of < 26
* History of other dementia-related neurological or psychiatric disorders, including psychotic developmental disorders, mania, depression, and schizophrenia
* Central neural system diseases, including traumatic brain injury, intracranial hemorrhage, and acute cerebral infarction
* Acute complications of diabetes, including diabetic ketoacidosis, hyperglycemic hyperosmolar state, and hypoglycemic coma
* Complicated with severe impairment of liver, kidney or heart function
* Metal implants, unable to complete the MR scanning
* Pregnant or lactating women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM patients will be recruited from the outpatient and inpatient units of the endocrinology department of the investigator's hospital. Healthy control will be recruited in the community
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-18 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Baseline cognitive performance | Day 1 of entry study
  The Montreal Cognitive Assessment (MoCA) score, ranges from 0 to 30, and higher scores mean better cognition.
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study and preserved at -81 °C in the Biobank of Drum Tower Hospital until examination.
  Aβ40, Aβ42, P-tau 181, P-tau 231, GFAP and NfL.
Baseline simultaneous EEG-fMRI | Within 1 week after cognitive assessments
  Frequency domain and spectrum domain analyses
Baseline brain structural MRI scan | Within 1 week after cognitive assessments
  Cortical morphology
Baseline brain functional MRI scan | Within 1 week after cognitive assessments
  Large-scale network functional connectivity

SECONDARY OUTCOMES:
Longitudinal changes of cognitive performance | From baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
  Compare the change of MoCA score from baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
Longitudinal changes of peripheral blood neuropathology biomarkers level | From baseline to final follow-up time points (36 months).
  Compare the changes of peripheral blood neuropathology biomarkers level from baseline to final follow-up time points (36 months).
Longitudinal changes of simultaneous EEG-fMRI | From baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
  Compare the change of frequency domain and spectrum domain from baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
Longitudinal changes of brain structural MRI scan | From baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
  Compare the changes of cortical morphology from baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
Longitudinal changes of brain functional MRI scan | From baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).
  Compare the changes of large-scale network functional connectivity from baseline to each follow-up time points (6 months, 12 months, 18 months, 24 months, 30months, 36 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be made during the 12 months after the end of study, and the original data can be obtained from the PI if necessary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: during the 12 months after the end of study